CLINICAL TRIAL: NCT05539898
Title: Improving the Criteria for Selecting Patients for Primary Prevention of Sudden Cardiac Death by Stratification of the Risk of Stable Ventricular Tachyarrhythmias
Brief Title: Improving the Criteria for Selecting Patients for Primary Prevention of Sudden Cardiac Death by Arrhythmic Risk Stratification
Acronym: PERFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Astrakhan Federal Centre For Cardiac Surgery (Other)
Responsible Party: Principal Investigator, Nikolay Ilov, Principal Investigator, Astrakhan Federal Centre For Cardiac Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ONRS_01
Record Dates: First submitted 2022-09-12; First posted 2022-09-14 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: sudden cardiac death; heart failure; primary prevention; risk stratification
MeSH Terms: conditions — Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICD (Other): ICD implanted
  Interventions: Device: ICD implantation

INTERVENTIONS:
Device: ICD implantation — All included in the study will undergo ICD implantation for primary prevention of SCD

SUMMARY:
A number of large randomized studies have demonstrated the importance of left ventricle ejection fraction (LV EF) for ventrucular tachyarhrythmia's (VT) prediction. The use of this indicator as the sole predictor of high arrhythmic risk requiring ICD implantation is enshrined in the current clinical recommendations. At the same time, many experts consider LV EF as too generalized indicator, which can be an integral indicator of total cardiovascular mortality, but lacks specificity in determining the risk of VT. It is known that only about 20% of patients with ICD implanted for primary prevention of sudden cardiac death (SCD) receive appropriate life-saving therapy.

Purpose of the study: to develop additional criteria for selection of patients with heart failure for implantation of cardioverter-defibrillator for the purpose of primary SCD prevention on the basis of stratification of the risk of occurrence of stable ventricular tachyarrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* LV EF ≤ 35% inspite of optimal drug therapy of heart failure (3 months and longer)
* NYHA II-IV
* favorable prediction of survival for 1 year or more

Exclusion Criteria:

* secondary SCD prevention
* indications for open heart surgery
* hypertrophic cardiomyopathy
* arrhythmogenic right ventricular dysplasia
* genetic channelopathies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 450 (Estimated)
Dates: Start 2017-01-13 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-12-29 (Estimated)

PRIMARY OUTCOMES:
Rate of VT primary occurrence | 24 months
  A stable paroxysm of VT (lasting ≥ 30 seconds) detected in the "monitoring" zone of VT, or paroxysm of VT, requiring ICD therapy.

SECONDARY OUTCOMES:
Rate of Cardiac Mortality | 24 months
  Registration of cardiac death
Number of Participants with CRT Response | 24 months
  Registration of CRT Response evaluated by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Federal Center for Cardiovascular Surgery, Astrakhan, Astrakhan Oblast, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ilov NN, Palnikova OV, Stompel DR, Nechepurenko capital A, CyrillicA. Clinical Predictors of Occurrence of Ventricular Tachyarrhythmias in Patients with Reduced Left Ventricle Ejection Fraction. Results of Single-Center Prospective Study. Kardiologiia. 2021 May 31;61(5):32-40. doi: 10.18087/cardio.2021.5.n1480. English, Russian. PMID 34112073